CLINICAL TRIAL: NCT03841825
Title: Effects of Active Reminders and Motivational Techniques on Oral Hygiene and Gingival Health in Orthodontic Patients: a Randomized Clinical Trial
Brief Title: Effects of Active Reminders and Motivational Techniques on Oral Hygiene and Gingival Health in Orthodontic Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: HM20014910
Record Dates: First submitted 2019-02-12; First posted 2019-02-15 (Actual); Last update posted 2020-09-10 (Actual); Status verified 2020-09

CONDITIONS: Oral Hygiene; White Spot Lesion; Gingivitis
MeSH Terms: conditions — Gingivitis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control (No Intervention): No messages or oral hygiene instructions
- Text message reminders (Experimental): Standardized text reminding patients to brush their teeth will be sent at 5:15 PM on Thursdays
  Interventions: Behavioral: Oral hygiene instructions
- In-person oral hygiene instructions (Active Comparator): Oral hygiene instructions and motivation during visit
  Interventions: Behavioral: Oral hygiene instructions
- Text messages and in-person instructions (Experimental): standardized text reminding patients to brush their teeth will be sent at 5:15 PM on Thursdays and oral hygiene instructions and motivation during visit
  Interventions: Behavioral: Oral hygiene instructions

INTERVENTIONS:
Behavioral: Oral hygiene instructions — Oral hygiene instructions and motivation
  Arms: In-person oral hygiene instructions; Text message reminders; Text messages and in-person instructions

SUMMARY:
This study will compare the use of text message reminders versus multiple in-person sessions of oral hygiene instructions and motivation on improving oral hygiene measurements.

DETAILED DESCRIPTION:
Orthodontic treatment (i.e. braces) makes it hard to keep good oral hygiene. The purpose of this research study is to compare the use of text message reminders versus multiple in-person sessions of oral hygiene instructions and motivation on improving oral hygiene measurements. Participation in this study will last up to 6 months and will consist of 4 study visits to the VCU Orthodontic clinic which are also regular visits for treatment. Measurements to assess participant's oral health will be taken during these visits. Participants will be randomly assigned to 1 of 4 groups which may include receiving different types of text messages, repeated in-person oral hygiene instructions, or both, or neither.

ELIGIBILITY:
Inclusion Criteria:

1. Age 11-20 that have their own mobile device
2. Patients have cellular plan that allows them to receive text messages at no extra cost
3. Patients that will undergo treatment with full fixed appliances

Exclusion Criteria:

1. patients with significant medical or dental history, including patients with bleeding disorders that would require antibiotic prophylaxis
2. Pregnant women

Ages: 11 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 67 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2020-03-06 (Actual); Study Completion 2020-03-06 (Actual)

PRIMARY OUTCOMES:
Change in 3-item Bleeding Index (BI) | Initial visit to 4 - 6 weeks
  Dental examiner observation of gum bleeding during exam after wires have been removed and participant has brushed teeth. Ratings are 0=absence of bleeding after 30 seconds, 1=bleeding observed after 30 seconds, 2=immediate bleeding
Change in 3-item Bleeding Index (BI) | 4 - 6 weeks to 8 - 12 weeks
  Dental examiner observation of gum bleeding during exam after wires have been removed and participant has brushed teeth. Ratings are 0=absence of bleeding after 30 seconds, 1=bleeding observed after 30 seconds, 2=immediate bleeding
Change in 3-item Bleeding Index (BI) | 8 - 12 weeks to 12 - 18 weeks
  Dental examiner observation of gum bleeding during exam after wires have been removed and participant has brushed teeth. Ratings are 0=absence of bleeding after 30 seconds, 1=bleeding observed after 30 seconds, 2=immediate bleeding

SECONDARY OUTCOMES:
Change in 5-item Modified Gingival Index (MGI) | Initial visit to 4 - 6 weeks
  Dental examiner observation of inflammation during exam after wires have been removed and participant has brushed teeth. Ratings are 0=Absence of inflammation, 1=Mild inflammation (marginal or papillary unit), 2=Mild inflammation (entire marginal and papillary unit), 3=Moderate inflammation, 4=severe inflammation
Change in 5-item Modified Gingival Index (MGI) | 4 - 6 weeks to 8 - 12 weeks
  Dental examiner observation of inflammation during exam after wires have been removed and participant has brushed teeth. Ratings are 0=Absence of inflammation, 1=Mild inflammation (marginal or papillary unit), 2=Mild inflammation (entire marginal and papillary unit), 3=Moderate inflammation, 4=severe inflammation
Change in 5-item Modified Gingival Index (MGI) | 8 - 12 weeks to 12 - 18 weeks
  Dental examiner observation of inflammation during exam after wires have been removed and participant has brushed teeth. Ratings are 0=Absence of inflammation, 1=Mild inflammation (marginal or papillary unit), 2=Mild inflammation (entire marginal and papillary unit), 3=Moderate inflammation, 4=severe inflammation
Change in 6 item Plaque index (PI) | Initial visit to 4 - 6 weeks
  Dental examiner observation of plaque during exam after wires have been removed and participant has brushed teeth. Ratings are 0= no plaque, 1=Discontinuous band of plaque at gingival margin, 2=Up to 1-mm continuous band of plaque at gingival margin, 3=Band of plaque wider than 1 mm but less than 1/3 of surface, 4=Plaque covering between 1/3 and 2/3 of surface, 5=Plaque covering 2/3 or more of surface
Change in 6 item Plaque index (PI) | 4 - 6 weeks to 8 - 12 weeks
  Dental examiner observation of plaque during exam after wires have been removed and participant has brushed teeth. Ratings are 0= no plaque, 1=Discontinuous band of plaque at gingival margin, 2=Up to 1-mm continuous band of plaque at gingival margin, 3=Band of plaque wider than 1 mm but less than 1/3 of surface, 4=Plaque covering between 1/3 and 2/3 of surface, 5=Plaque covering 2/3 or more of surface
Change in 6 item Plaque index (PI) | 8 - 12 weeks to 12 - 18 weeks
  Dental examiner observation of plaque during exam after wires have been removed and participant has brushed teeth. Ratings are 0= no plaque, 1=Discontinuous band of plaque at gingival margin, 2=Up to 1-mm continuous band of plaque at gingival margin, 3=Band of plaque wider than 1 mm but less than 1/3 of surface, 4=Plaque covering between 1/3 and 2/3 of surface, 5=Plaque covering 2/3 or more of surface

CONTACTS AND LOCATIONS:
Overall Officials: Shroff Bhavna, DDS, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No